CLINICAL TRIAL: NCT06118320
Title: The Clinical Study Utilizing Gut Microbiota and Metabolomics to Investigate the Efficacy of Potassium Sodium Hydrogen Citrate Therapy in the Treatment of Uric Acid Kidney Stones.
Brief Title: The Effective of Potassium Sodium Hydrogen Citrate in Treating Uric Acid Stones Using Gut Microbiota and Metabolomics.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cheng Cao (Other)
Responsible Party: Sponsor-Investigator, Cheng Cao, MD, Changshu Affiliated Hospital of Soochow University
Organization: Changshu Affiliated Hospital of Soochow University (Other)
Other Study IDs: ChangshuAHSU
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Uric Acid Stones
Keywords: gut microbiota; renal uric acid stone; 16S rRNA; short chain fatty acid; potassium sodium hydrogen citrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug treatment group of uric acid stones（DT group）: Potassium sodium hydrogen citrate granules (MADAUS GMBH, Germany, 2.5g/packet) were administered to patients with residual stones (>5 mm in diameter) after surgery or difficult-to-remove stones in the infrarenal calyces for a three-month intervention period. The medication was taken as follows: one packet after breakfast, one packet after lunch, and two packets after dinner. Participants were instructed to abstain from alcohol consumption, smoking, and the use of any probiotics or medications that lower uric acid levels during the therapeutic period.They were also instructed to monitor preprandial urine pH levels to maintain an effective range of 6.2-6.8.
  Interventions: Drug: Potassium sodium hydrogen citrate

INTERVENTIONS:
Drug: Potassium sodium hydrogen citrate — Medication: Potassium sodium hydrogen citrate granules (MADAUS GMBH, Germany, 2.5g/package).
  Method: Preprandial urine pH was monitored to maintain an effective range of 6.2 to 6.8. One package should be taken after breakfast, one after lunch, and two after dinner. If the pH falls below 6.2, a half-package dose should be added; if it exceeds 6.8, a half-package dose should be reduced accordingly. Oral medication will be administered for a duration of three months.
  Medication requirements: Abstain from alcohol and smoking during treatment period and avoid using any probiotics or drugs that lower uric acid levels.
  Other Names: PSHC

SUMMARY:
The goal of this observational study is to investigate the alterations in gut microbiota and metabolites among patients with uric acid stones following the administration of potassium sodium hydrogen citrate. The main question it aims to predict the potential metabolic mechanism and therapeutic target of potassium sodium hydrogen citrate in treating uric acid stones through analysis of gut microbiota and metabolomics. The participants were required to undergo a 3-month drug intervention, providing blood, urine, and stool samples before and after treatment. No additional interventions were implemented for the subjects.

DETAILED DESCRIPTION:
The objectives of this study were to investigate the association between the presence of bacterial genera and short-chain fatty acids (SCFAs) in stool, as well as biochemical elements in blood and urine, among patients with uric acid nephrolithiasis. The sensitivity difference of potassium sodium hydrogen citrate in treating uric acid kidney stones was examined through gut microbiota analysis and metabolomics to predict potential metabolic mechanisms and sensitive targets for treatment. Blood biochemistry, 24-hour urine composition analysis, and other indicators were collected from the subjects. Fecal samples were obtained for 16S ribosomal RNA sequencing to analyze the characteristics of gut microbiota in relation to blood and urine biochemical metabolism indicators. Subjects received treatment with potassium sodium hydrogen citrate granules for a duration of 3 months. Blood and urine biochemical indexes, fecal samples, 16S ribosomal RNA sequencing data, and short-chain fatty acid levels in fecal samples were collected before and after treatment. The care of the enrolled patients will not be subject to any intervention.

ELIGIBILITY:
Inclusion Criteria:

All stone patients were diagnosed using urologic ultrasonography, kidney-ureter-bladder (KUB) X-ray, or abdominal computed tomography (CT). Stone samples were obtained through ureteroscopic lithotripsy (URSL), percutaneous nephrolithotomy (PCNL), or extracorporeal shock wave lithotripsy (ESWL). Stones were analyzed using an automated infrared spectroscopy system, LIIR-20 (Lanmode Scientific Instrument Co., Ltd., Tianjin, China), and the main components were determined based on the most abundant substances listed in the report, which were classified as pure or mixed uric acid stones (anhydrous uric acid content >50%).

Exclusion Criteria:

Patients with malignancy, chronic liver insufficiency, a history of statin use, and thyroid or parathyroid disease were excluded from the study. Similarly, individuals with a history of urolithiasis or dyslipidemia as well as those who had used statins were excluded from the control group. Participants were also excluded if they had taken antibiotics or immune suppressants within one month prior to fecal sampling, or had a history of chronic diarrhea or constipation, chronic enteritis, irritable bowel syndrome, gastrointestinal tumors or intestinal surgery.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stone patients were diagnosed using urologic ultrasonography, kidney-ureter-bladder (KUB) X-ray, or abdominal computed tomography (CT). Stone samples were obtained through ureteroscopic lithotripsy (URSL), percutaneous nephrolithotomy (PCNL), or extracorporeal shock wave lithotripsy (ESWL). Stones were analyzed using an automated infrared spectroscopy system, LIIR-20 (Lanmode Scientific Instrument Co., Ltd., Tianjin, China), and the main components were determined based on the most abundant substances listed in the report, which were classified as pure or mixed uric acid stones (anhydrous uric acid content >50%).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum diameter of stone | From enrollment to the end of treatment at 3 months
  The patients underwent pre- and post-drug intervention abdominal CT examinations, enabling determination of the stone's maximum diameter（mm） through analysis of CT images.
Gut microbiota analysis | From enrollment to the end of treatment at 3 months
  The fecal samples were collected pre- and post-intervention for the analysis of gut microbiota.
Short chain fatty acid contents | From enrollment to the end of treatment at 3 months
  The collection of fecal samples was conducted both pre- and post-intervention in order to assess the levels of short-chain fatty acids.

SECONDARY OUTCOMES:
Serum triglycerides | From enrollment to the end of treatment at 3 months
  The peripheral venous blood was collected pre- and post-intervention, and the serum triglyceride level (mmol/L) was measured by automatic biochemical analyzer.
Serum cholesterol | From enrollment to the end of treatment at 3 months
  The peripheral venous blood was collected pre- and post-intervention, and the serum cholesterol level (mmol/L) was measured by automatic biochemical analyzer.
Serum high density lipoprotein cholesterol | From enrollment to the end of treatment at 3 months
  The peripheral venous blood was collected pre- and post-intervention, and the serum high density lipoprotein cholesterol level (mmol/L) was measured by automatic biochemical analyzer.
Serum low density lipoprotein cholesterol | From enrollment to the end of treatment at 3 months
  The peripheral venous blood was collected pre- and post-intervention, and the serum low density lipoprotein cholesterol level (mmol/L) was measured by automatic biochemical analyzer.
Serum creatinine | From enrollment to the end of treatment at 3 months
  The peripheral venous blood samples were collected from the subjects both before and after the intervention, and the serum creatinine levels（μmol/L） were measured by automatic biochemical analyzer.
Serum uric acid | From enrollment to the end of treatment at 3 months
  The peripheral venous blood samples were collected from the subjects both before and after the intervention, and the serum uric acid levels（μmol/L） were measured by automatic biochemical analyzer.
Serum potassium | From enrollment to the end of treatment at 3 months
  The peripheral venous blood samples were collected from the subjects both before and after the intervention, and the serum potassium levels（mmol/L） were measured by automatic biochemical analyzer.
Serum magnesium | From enrollment to the end of treatment at 3 months
  The peripheral venous blood samples were collected from the subjects both before and after the intervention, and the serum magnesium levels（mmol/L） were measured by automatic biochemical analyzer.
Urine pH | From enrollment to the end of treatment at 3 months
  The urine pH value was assessed by collecting mid-stream urine samples before and after the intervention by automatic biochemical analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Cao, MD, Principal Investigator — The Changshu Hospital Affiliated to Soochow University
Locations (1):
- Changshu Hospital Affiliated to Soochow University, Changshu, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No